CLINICAL TRIAL: NCT05114668
Title: A Phase 1, First-in-Human, Open-Label Study to Assess the Safety, Tolerability, and Pharmacokinetics of EVT801 in Patients With Advanced Solid Tumours
Brief Title: Safety, Tolerability, and Pharmacokinetics of EVT801 in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kazia Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KZA-0801-101
Record Dates: First submitted 2021-10-06; First posted 2021-11-10 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumor, Adult
Keywords: cancer; solid tumors; advanced or metastatic tumors; renal cell carcinoma; soft tissue sarcoma
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Carcinoma, Renal Cell; Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stage 1 (Experimental): - Stage 1 (Dose Escalation Cohorts): Stage 1 is a multiple ascending dose escalation of EVT801 in patients with advanced solid tumours to evaluate the safety and tolerability of EVT801 and to determine MTD / RP2D for further investigation.
  Interventions: Drug: EVT801
- Stage 2 (Experimental): - Stage 2 (Biomarker Expansion cohorts): A biomarker expansion cohort, in which all subjects will receive EVT801 at the MTD / RP2D, will be recruited to explore pharmacodynamic outcomes and further elucidate tolerability, activity, and pharmacokinetics.
  Interventions: Drug: EVT801

INTERVENTIONS:
Drug: EVT801 — Stage 1: Patients will be dosed orally with EVT801 capsules at the dose and schedule to which they are assigned.
  Stage 2: Patients will be dosed orally with EVT801 capsules at the MTD / RP2D identified in Stage 1 of the study.

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of EVT801 in subjects with advanced or metastatic solid tumours. The study also aims to determine the maximum tolerated dose (MTD) and / or a recommended Phase 2 dose (RP2D) of EVT801 when administered daily to subjects with advanced or metastatic solid tumours.

The study comprises two stages, each with distinct purposes, patient populations, and procedures:

* Stage 1: a multiple ascending dose escalation of EVT801 to evaluate the safety and tolerability of EVT801 and to determine MTD / RP2D in subjects with advanced solid tumours.
* Stage 2: a biomarker expansion cohort, in which all subjects will receive EVT801 at the MTD / RP2D, to explore pharmacodynamic outcomes and further elucidate tolerability, activity, and pharmacokinetics.

DETAILED DESCRIPTION:
Stage 1 - Dose Escalation Cohorts:

Stage 1 is a multiple ascending dose escalation of EVT801 in patients with advanced solid tumours to determine MTD / RP2D for further investigation.

After completing screening and signing informed consent, subjects will be enrolled. The first dose of study drug will be administered at the site, and patients will undergo intensive PK assessment for 48 hours before receiving the second and subsequent doses.

The first subject in Stage 1 will receive EVT801 at a dose of 50 mg QD (Quaque Die: once daily) (Dose Level 1). If no Doses Limiting Toxicity (DLTs) are observed in a 28-day period, the second subject may be enrolled at Dose Level 2. The study will proceed by way of single-patient cohorts until (a) treatment-related toxicity of at least Grade 2 is observed, or (b) Dose Level 5 is reached, or (c) the Principal Investigator, in consultation with the sponsor, determines that it is appropriate to transition to larger cohorts. At this point, the study will move to a conventional 3+3 design.

If a DLT is observed in any cohort, that cohort will expand to six patients. If two DLTs are observed at a given dose level, the prior dose level will be declared the MTD, and Stage 1 will be deemed complete. If the prior dose level had recruited only a single patient, then that dose level will be expanded to three patients, such that the MTD will have been administered to a minimum of three patients.

If two DLTs are observed at Dose Level 2 (100 mg QD), a de-escalation cohort (Dose Level -1) will enrol three patients in order to establish the viability of twice-daily dosing.

Once the MTD has been established, the sponsor will evaluate, in consultation with the investigators, whether that dose or a lower dose should be used for subsequent investigation (the RP2D). This evaluation will be based on a consideration of broader factors than safety, including PK and PD. The RP2D shall under no circumstances be greater than the MTD.

The sequence of doses examined will be:

50 mg QD → 100 mg QD (→50 mg BID [Bis In Die (i.e. twice daily)] if 2 DLTs / 6 patients @ 100 mg QD) → 100 mg BID → 200 mg BID → 400 mg BID → 500 mg BID → 600 mg BID → 800 mg BID (up to 8 cohorts).

After completion of at least two cycles at the dose level to which they were initially assigned, individual subjects may escalate to higher dose levels, providing the higher dose level has (a) been administered to at least one patient for at least 28 days without grade 2 treatment-related toxicity, or (b) been administered to at least three subjects for at least 28 days without a DLT, or (c) been administered to at least six subjects for at least 28 days with no more than one DLT. A given subject may escalate through multiple dose levels in this fashion, providing the aforementioned criteria continue to be satisfied and the patient has no ongoing clinically significant adverse event > grade 1.

Stage 2 - Biomarker Expansion Cohorts:

Immediately following determination of the MTD / RP2D in Stage 1, Stage 2 will open to recruitment.

Stage 2 comprises two sub-components:

* Stage 2A :patients with advanced renal cell carcinoma.
* Stage 2B: patients with advanced soft-tissue sarcoma. Subjects may be enrolled in parallel, as they become available through screening.

All subjects in Stage 2 will receive EVT801 at the MTD / RP2D established in Stage 1.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of any gender who are ≥18 years of age at the time of study entry.
2. Histologically-confirmed advanced or metastatic solid tumours, unresponsive to standard treatment, or for whom no standard treatment is available or appropriate.
3. Measurable or evaluable disease per RECIST 1.1 criteria.
4. ECOG performance status <2.
5. Life expectancy of greater than 3 months, in the opinion of the investigator.
6. Able and willing to provide archived tumour samples, or to undergo pre-treatment tumour biopsy if feasible; subjects must be able to provide at least one tumour tissue sample (archived or pre-treatment biopsy) to be eligible.
7. Written, signed, and dated informed consent to participate in this study in a format approved by the ethics committee.
8. Adequate organ and bone marrow function at the time of screening, including:

   Haematology:
   * Absolute neutrophil count (ANC) >1.5 x 109/L.
   * Platelet count of >75 x 109/L.
   * Haemoglobin > 90g/L (without transfusion for at least 2 weeks).

   Renal Function:
   * Estimated glomerular filtration rate (GFR), based on MDRD (modification of diet in renal disease) calculation, of ≥60 ml/min/1.73 m2.
   * Creatinine ≤1.5 mg/dL (≤132.6 μmol/L).
   * Urine dipstick for proteinuria <2+. Subjects discovered to have ≥2+ proteinuria on dipstick urinalysis should undergo a 24-hour urine collection and must demonstrate ≤1.0 g of protein in 24 hours OR Urine protein/creatinine ratio ≤1.0.

   Liver Function:
   * Total bilirubin ≤1.5 x ULN (<2 x ULN for subjects with suspected Gilbert's syndrome).
   * AST and ALT <2.5 x ULN (<5 x ULN if liver metastases are present).
   * Alkaline phosphatase <3 x ULN (<5 x ULN if liver or bone metastases are present).

   Coagulation:
   * Prothrombin time (PT) <1.5 x ULN.
   * Partial thromboplastin time (PTT) <1.5 x ULN.
   * International normalised ratio (INR) <1.5 x ULN (or within target range if on prophylactic anticoagulation therapy).
9. The effects of EVT801 on the developing human foetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (e.g. hormonal or barrier method of birth control) prior to study entry and for the duration of study participation and for a period of 6 months after the last dose of study medication; female subjects will be required to demonstrate a negative serum pregnancy test prior to study entry and subjects who are lactating should be excluded. Fertile men (as defined in section 5.5) must agree to use adequate contraception up to 90 days after the last dose of EVT801 according to the latest version of the CTFG Contraception Guidance.
10. Able and willing, in the judgment of the investigator, to meet all protocol-required treatments, investigations and visits. This must include the ability for the subject to comply with daily self-administration of an oral therapy, or reliable means for treatment to be administered by a dependable third party such as a relative or caregiver. Subjects must also be able and willing to undergo magnetic resonance imaging, and to receive gadolinium-containing contrast media.

Additional Inclusion Criteria for Stage 2:

1. Subjects with a histologically confirmed diagnosis of advanced renal cell carcinoma (Stage 2A) or advanced soft tissue sarcoma (Stage 2B).
2. Subjects who are suitable and willing to provide two biopsies of tumour tissue (pre-treatment and on-treatment).

Exclusion Criteria:

1. Recent history of antitumor therapy administered with the intent of treating cancer prior to study entry, including pharmacological agents, surgical procedures, or radiotherapy; symptomatic treatments such as analgesia or steroids are permitted; palliative radiotherapy is permitted, providing it is completed at least two weeks prior to study entry. Exclusion period will be adapted to the previous line of therapy: 6 weeks for nitrogen mustard type alkylating agents, 4 weeks for monoclonal antibodies, 3 weeks for standard chemotherapy and 2 weeks or 5 half-lives for small molecule targeted agents and hormonal therapy.
2. Any unresolved toxicity from prior treatment of Grade ≥2, according to NCI CTCAE version 5.0, except for alopecia, vitiligo, supplemented and stable endocrine disorders following immuno-oncology treatment or abnormal laboratory parameters within the ranges defined in the inclusion criteria.

   Subjects with Grade ≥2 neuropathy, and subjects with irreversible toxicity that is not reasonably expected to be exacerbated by study participation, may be included only after consultation with the lead investigator.
3. CNS tumours: symptomatic or steroid-dependent lesions. Cured lesions are acceptable.
4. History of another primary malignancy, unless treated with curative intent and with no known active disease for ≥2 years prior to study entry; subjects with a history of adequately treated non-melanoma skin cancer or superficial bladder cancer or carcinoma in situ of the cervix may be enrolled if there is no evidence of residual disease.
5. Current participation in another interventional clinical trial, or participation within 28 days prior to study entry.
6. Clinically significant cardiac disease or impaired cardiac function, including:

   * Congestive heart failure requiring treatment (New York Heart Association (NYHA) Grade ≥2).
   * Left ventricular ejection fraction (LVEF) <50%, as determined by MUGA scan or echocardiogram.
   * History or current evidence of clinically significant or uncontrolled cardiac arrhythmias, atrial fibrillation, or conduction abnormality.
   * Acute coronary syndromes, myocardial infarction, unstable angina, or procedures including coronary artery bypass grafting (CABG) or coronary angioplasty within 6 months prior to screening.
   * Uncontrolled hyperkalemia.
   * Mean (based on mean value of screening triplicate ECGs) resting corrected QT interval (QTc) > 470 msec (for women) and > 450 msec (for men) obtained from 3 consecutive ECGs or with QT interval > 500 msec for one of the ECGs at screening visit and D1 predose.
7. Any disease of the GI tract which renders the subject unable to take oral medications, or which might affect the absorption of oral medicines (e.g. inflammatory bowel disease, malabsorption syndrome, requirement for parenteral nutrition).
8. Active haemorrhagic syndrome, or presence of tumour in contact with large vessels (e.g. neck, mediastinum, retroperitoneum).
9. Acute infection within 1 week prior to starting study treatment.
10. Diagnosis of SARS-CoV-2, confirmed by PCR within 3 months prior to starting study treatment, unless fully resolved with no residual symptoms.
11. Known active infection including hepatitis B (HbsAg positive), hepatitis C, or HIV are not eligible; subjects with treated HBV or HCV infection with negative or stable PCR for HBV or HCV RNA are eligible; subjects with resolved HBV infection (anti-HBc positive and HBsAg negative) are eligible; subjects with HCV antibodies are eligible if negative PCR for HCV RNA.
12. Any pre-existing or intercurrent illness or pathology which, in the judgment of the investigator, has the potential to increase the safety risk associated with EVT801 administration, or to confound the results of the study.
13. History of severe allergic reactions to any unknown allergens or to any components of the study drug or to any other VEGFR3 inhibitor.
14. Subjects receiving any medications or substances that are moderate and/or potent CYP3A4 inhibitors which may have an effect on the metabolism of EVT801 should be excluded.
15. Subjects not covered by a healthcare insurance system.
16. Subjects deprived of liberty by a judicial or administrative decision, patient admitted to a social institution or who is under a measure of legal protection, patient hospitalized without consent or who is in an emergency situation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
MTD and / or a RP2D of EVT801 when administered daily to subjects with advanced or metastatic solid tumours. | 24 months
  The MTD is defined as the highest dose administered at which fewer than one-third of patients experienced a DLT.
  The RP2D will be determined for Stage 1 on the basis of an overall assessment of safety, pharmacokinetics, and other information. The RP2D may be equal to, or lower than, the MTD.
Adverse event (AE) safety information for EVT801 | 36 months
  To provide safety information for EVT801 by assessing adverse events, per CTCAE v5.0.

SECONDARY OUTCOMES:
Cmax pharmacokinetic (PK) parameter of EVT801 following administration in an oral capsule formulation. | 12 months
Tmax pharmacokinetic (PK) parameter of EVT801 following administration in an oral capsule formulation. | 12 months
T1/2 pharmacokinetic (PK) parameter of EVT801 following administration in an oral capsule formulation. | 12 months
AUC(0-last) and AUC(0-inf) pharmacokinetic (PK) parameter of EVT801 following administration in an oral capsule formulation. | 12 months
CL pharmacokinetic (PK) parameter of EVT801 following administration in an oral capsule formulation. | 12 months
Preliminary anti-tumour activity of EVT801 via assessment of overall response rate (ORR). | 36 months
  ORR will be defined as the proportion of patients in a given analysis population that demonstrate a best overall response of Complete Response (CR) or Partial Response (PR), based on investigator assessment using RECIST (v1.1) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Gomez-Roca, MD, Principal Investigator — Institut Claudius Regaud, Toulouse, France
Locations (2):
- France (2):
  - Centre Léon Bérard, Lyon
  - Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse